CLINICAL TRIAL: NCT02546115
Title: Assessing the Benefits of the Use of a Tension Night Splint in Patients With Plantar Fasciitis, a Single-blinded Randomised Controlled Trial
Brief Title: RCT - Assessing the Benefits of the Use of a Tension Night Splint in Patients With Plantar Fasciitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UHL - 11335
Record Dates: First submitted 2015-06-15; First posted 2015-09-10 (Estimated); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Plantar Fasciitis
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Intervention (Active Comparator): standard practice (structured rehabilitation programme) + TNS
  Interventions: Device: tension night splint; Other: standard practice - a structured rehabilitation programme
- control (Active Comparator): standard practice (structured rehabilitation programme)
  Interventions: Other: standard practice - a structured rehabilitation programme

INTERVENTIONS:
Device: tension night splint — this is the use of a commercially available tension night splint device, to be worn by the patient
  Arms: Intervention
Other: standard practice - a structured rehabilitation programme — this is the standardised structured rehabilitation programme of home exercises given to patients, with supporting literature, and instructions on how to progress the regime themselves

SUMMARY:
To assess whether the provision of a tension night splint (TNS) device has any additional benefit in patients with chronic plantar fasciitis, compared to routine care comprising physiotherapy & podiatry alone.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age >18 with symptoms of plantar fasciitis for >3 months
2. Diagnostic imaging confirming plantar fasciitis (either US or MRI acceptable)

Exclusion Criteria:

1. Current or previous partial or full-thickness tear of the Achilles tendon or plantar fascia (either clinically suspected or proven on imaging)
2. Current or previous calf muscle injury
3. Previous use of tension night splint
4. Diabetic neuropathy, or other sensory / sensorimotor disturbance
5. Lower limb vascular compromise
6. Fragile skin, or skin wounds on lower leg
7. Subjects with impaired mobility which prevents safe and effective application of the Tension Night Splint
8. Any other condition which it is thought may be aggravated by the use of a tension night splint
9. Subjects unable to give valid consent for the study
10. Subjects who state that they are unable or unwilling to undergo the home-based structured rehabilitation programme as a part of the study process
11. Subjects who are unable to attend the follow-up appointment required at the end of the study

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-09; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Reduction in pain as assessed by a 0-10 visual analogue scale (VAS) | primary outcome time = 3 months

SECONDARY OUTCOMES:
improvement in function as assessed by validated PROMs as described below | 3 months - end point
  several validated Patient rated Outcome Measures (PROMS) are used in this study, including: FFI-r, FAAM, and MOXFQ

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Wheeler, Principal Investigator — UHL
Locations (1):
- University Hospitals of Leicester NHS Trust, Leicester, United Kingdom

REFERENCES:
- [Derived] Wheeler PC. The addition of a tension night splint to a structured home rehabilitation programme in patients with chronic plantar fasciitis does not lead to significant additional benefits in either pain, function or flexibility: a single-blinded randomised controlled trial. BMJ Open Sport Exerc Med. 2017 Jun 13;3(1):e000234. doi: 10.1136/bmjsem-2017-000234. eCollection 2017. PMID 29259809
- See also: publication - open access — http://bmjopensem.bmj.com/content/3/1/e000234